CLINICAL TRIAL: NCT05577884
Title: Noise Reduction and Image Quality Improvement in Ultra-low-dose Whole-body CT Scans Using AI-based CT Reconstruction Program (ClariCT.AI) in Patients With Multiple Myeloma: A Prospective, Single-center Study
Brief Title: Ultra-low-dose Whole-body CT Using AI-based CT Reconstruction in Patients With Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Dong Chae, Clinical Professor, Seoul National University Hospital
Other Study IDs: SNUH-2021-4317
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Multiple myeloma: Patients with suspicion of multiple myeloma and scheduled for CT
  Interventions: Diagnostic Test: noncontrast-enhanced whole-body CT

INTERVENTIONS:
Diagnostic Test: noncontrast-enhanced whole-body CT — noncontrast-enhanced low-dose whole-body CT using dual-source CT scanner using A-tube (75% radiation) and B-tube (25% radiation).
  * conventional low-dose CT data (A +B tubes, 100% dose) are reconstructed with iterative reconstruction
  * ultra-low dose CT data (B-tube only, 25% dose) are reconstructed with deep learning commercially available software.

SUMMARY:
This prospective study aims to perform intra-individual comparison of the image quality between ultra-low-dose whole-body CT with deep learning reconstruction and conventional low-dose whole-body CT with iterative reconstruction in patients with suspected multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients with suspected multiple myeloma and scheduled for noncontrast-enhanced low-dose whole-body CT
* patients who have no previous history of chemotherapy for multiple myeloma

Exclusion Criteria:

* patients who do not agree to the protocol
* non-Korean patients
* pregnancy

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred to Hemoatooncology department with suspicion of multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Contrast-to-noise ratio | 3 months after the CT scan
  Contrast-to-noise ratio (CNR) of the vertebral body and paraspinal muscle obtained at L1 vertebra level

OTHER OUTCOMES:
Noise | 3 months after the CT scan
  Noise at paraspinal muscle
Signal-to-noise ratio (SNR) | 3 months after the CT scan
  Signal-to-noise ratio (SNR) at paraspinal muscle
Edge rising distance | 3 months after the CT scan
  Edge rising distance at vertebral cortex
Subjective overall image quality | 3 months after the CT scan
  Subjective overall image quality on four-point scale (1: worst, 4: excellent, representative value is average score)
Conspicuity of bone structure | 3 months after the CT scan
  Conspicuity of bone structure on four-point scale (1: worst, 4: excellent, representative value is average score)
Conspicuity of soft tissue | 3 months after the CT scan
  Conspicuity of soft tissue on four-point scale (1: worst, 4: excellent, representative value is average score)
Lesion detectability | 3 months after the CT scan
  Myeloma lesion detection rate on conventional low-dose CT and ultra-low-dose CT by blinded reviewers

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Dong Chae, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No